CLINICAL TRIAL: NCT04990713
Title: QORVATS Study. A Randomized Controlled, Triple Blinded to Compare the Quality of Recovery (QoR 40) Between Intercostal Block and a Combination of Intercostal Nerve Block With Serratus Plane Catheter for Patient's Undergoing VATS Procedures.
Brief Title: QoR40 Between Intercostal Block and Intercostal Block and Serratus Plane Catheter During VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Abhijit Biswas, Assistant Professor, Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QORVATS
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Video Assisted Thoracic Surgery (VATS); Pain Management
Keywords: Intercostal Block; Fascial Plane Block
MeSH Terms: conditions — Agnosia | interventions — Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: There will be two study groups. All study participants will receive serratus plane block (SAB) with catheter for continuous infusion and an intercostal block. Depending on the group allocation, the study participants may receive local anesthetics or placebo for the serratus plane block.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant, treating anesthesiologist and surgical team, and outcomes assessor will be blinded to prevent bias. One of the study team co-investigators who is not the treating anesthesiologist during the participants's surgery will prepare the study drugs. The treating anesthesiologist will not be aware of the contents of the study drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serratus Plane Block (Placebo) and Intercostal Block (Local Anesthestic) (Placebo Comparator): Patients randomized to this group will receive the intercostal block with local anesthetic and the serratus plane block with saline placebo. Local anesthetic administered will be ropivacaine 0.2%.
  Interventions: Procedure: Serratus Plane Block (Placebo) and Intercostal Block (Local Anesthestic)
- Serratus Plane Block (Local Anesthetic) and Intercostal Block (Local Anesthetic) (Experimental): Patients randomized to this group will receive the intercostal block with local anesthetic and the serratus plane block with local anesthetic. Local anesthetic administered will be ropivacaine 0.2%.
  Interventions: Procedure: Serratus Plane Block (Local Anesthetic) and Intercostal Block (Local Anesthetic)

INTERVENTIONS:
Procedure: Serratus Plane Block (Local Anesthetic) and Intercostal Block (Local Anesthetic) — Patients will receive local anesthetic via serratus plane block as opposed to saline placebo
  Other Names: Serratus Plane Block administering Ropivacaine 0.2%
  Arms: Serratus Plane Block (Local Anesthetic) and Intercostal Block (Local Anesthetic)
Procedure: Serratus Plane Block (Placebo) and Intercostal Block (Local Anesthestic) — Patients will receive saline placebo via serratus plane block
  Other Names: Serratus Plane Block administering Saline Placebo
  Arms: Serratus Plane Block (Placebo) and Intercostal Block (Local Anesthestic)

SUMMARY:
Video assisted thoracic surgery (VATS) has emerged as standard of care for majority of thoracic surgeries. It is less invasive compared to thoracotomy and is associated with improved perioperative outcomes [1-3]. Good perioperative analgesia after thoracic surgery will enable pulmonary toilet, early chest physiotherapy and mobilisation, [4,5,6]. Thirty-day hospital visits and hospital readmissions at London Health Sciences Centre (LHSC) is around 21% and 9% respectively [7]. One of the top five determinant for hospital visit and readmission in 30 days, was persistent post operative pain [7].

Several options to analgesia are available for patients undergoing VATS procedure. Systemic opioid based multimodal analgesia, central neuraxial blocks like thoracic epidural and peripheral nerve blocks are different available options, and their practise varies across institution [4,8,9]. Thoracic epidural or paravertebral blocks can be challenging to perform with high failure rates [10-12].

Fascial plane blocks (SAB; ESP) are in vogue in the present era [13-16]. They are easy to perform and do not require similar dexterity as needed to perform thoracic epidural or paravertebral blocks. They have minimal side effects and provide the options for continuous infusion for prolonged analgesia. They have become an effective part of multimodal analgesia and have established their roles in ERAS (enhanced recovery after surgery) protocol for VATS procedures.

SAB has become a common practise at our institution with proved clinical efficacy.

Perioperative Surgical Home is a patient centric team-based approach to improve patient's experiences in the perioperative period and thus improve healthcare [17]. Quality of Recovery (QoR) is a key determinant to perioperative surgical home and can be measured using the QoR 40 score [18]. This is a well validated score with a minimal important clinical difference (MICD) of 6.3 [19]. Quality of recovery combines five dimensions of health: patient support, comfort, emotions, physical independence and pain to achieve a single patient outcome - improved patient care [18].

The investigators hypothesize the that patients undergoing VATS lung resections using a combination of intercostal nerve block plus continuous SAB catheter infusion of local anesthetics will have a 20% increase in their QoR-40 score 24hour after the surgery compared to a single shot intercostal nerve block.

DETAILED DESCRIPTION:
This is a prospective randomized controlled triple-blind study. There will be two study groups. All study participants will receive SAB with catheter for continuous infusion and intercostal block. Depending on the group allocation, the study participants may receive local anesthetics or placebo for the block.

Participants depending on the group allocation, will either receive ropivacaine 0.2% or equal volume of normal saline (placebo) solutions for the nerve blocks. This is meant to maintain participant, clinical team, and investigator blinding. The anesthetist(s) performing the block will be blinded to the intervention along with the anesthetists performing the general anesthesia and the surgical team. Importantly, the intraoperative and postoperative opioids will be administered by anesthetists and nurses, respectively, who are blinded to group allocation. Furthermore, the research coordinator collecting all outcome data will also be blinded Interventions Intraoperative anesthetic managements will depend on the anesthesiologists in care of the patient on that day and will be based on standard of institutional practise and Canadian anesthesia society guidelines irrespective of patient study participation. Intraoperatively, the patient will receive Opioids or NSAIDS on discretion of the anesthesiologists depending on the clinical need. To standardize the perioperative multimodal analgesic management and to reduce biases, none of these patients will receive any ketamine or gabapentin during the perioperative period. All the study interventions will be performed after completion of surgery and when the patient is still under anesthesia. After the completion of surgery, with patient still on lateral decubitus, surgical site being non dependant, the thoracic wall will be cleaned with 2% chlorhexidine solution and draped aseptically to maintain a sterile environment. The intercostal block will be completed by the surgical team while the serratus catheter will be performed by one of the anesthesiologist coinvestigators. The study drugs will be prepared by a different co-investigator and the anesthesiologists performing the block or providing general anesthesia for the patient will not be aware of the content of the study drugs.

Patients will be recovered from anesthesia once the blocks are complete and transferred to PACU for recovery. All the patients will receive opioid based patient-controlled analgesia (PCA) with hydromorphone or morphine only along with acetaminophen in the postoperative period. These are standard of care at LHSC. The participants will also receive 0.2% ropivacaine infusion 7 mL/hr or normal saline infusion 7mL/hr depending on the study group. Their postoperative pain will be managed by the acute pain services as per standard hospital guidelines irrespective of their study participation.

One of the study team members will access the patient in the postoperative period (PACU and once daily) until discharge for data collection.

Intercostal nerve block The intercostal block will be performed by the surgical team under direct vision using thoracoscope. 5 mL of 0.2% ropivacaine will be injected at each 4th,5th,6th and 7thintercostal nerve at posterior axillary line. After full asepsis and placement of thoracoscope respective ribs will be palpated to identify the inferior border and neuronal anatomy will be identified using video assistance thoracoscope. Study drugs will be injected at the inferior border at midaxillary line at each space. Total volume of study drugs injected will be 20 mL.

SAB catheter The ultrasound (Sonosite) transducer will be placed in a caudal to cranial orientation on the mid axillary line at the level of the 5th rib. The target fascial plane between the serratus anterior (superficial) and the external intercostal (deep) muscles and the rib will be identified, and the path of the block needle will be determined. Braun, contiplex Touhy ultra echogenic needle with non stimulating catheter system for continuous nerve will be used. The needle will be inserted at the cranial aspect of the ultrasound probe and advanced in-plane to target the fascial plane directly below the serratus muscle. Once the tip is verified in the correct position, 10 mL of 0.2% ropivacaine or normal saline will be injected into the plane slowly in 5 mL aliquots under frequent aspiration and correct spread in the interfacial plane will be observed. The catheter will be placed in the plane and another 10 mL of 0.2% ropivacaine or normal saline will be injected through the catheter to verify the catheter placement.

Sample size calculation Sample size calculations were based on the study published by Do-Hyeong Kim et al [15] The calculation for the projected sample size is as follows. For MCID(minimal clinically important difference)- 6.3; Beta = 80% power, alpha = 0.05 N = 7.85 x [ (14.4)2 + (15.9)2] / (6.3)2 = 7.85 x [207.36 + 252.81] / 39.69 = 91 Sample size for one group = 91 Sample size for two groups = (91x2) = 182 Sample size for 10% loss in follow-up = 200 (approximately 100 in each group)

Statistical Analysis Baseline data will be presented in tabular form by treatment group. Categorical variables will be summarized as number (%). Percentages will be calculated according to the number of patients for whom data is available. Where values are missing, the denominator will be stated in the Table. Normality of continuous outcomes will be assessed visually (using histograms of raw and/or transformed data) and numerically (using the Shapiro-Wilk test). If the raw or transformed data are approximately normally-distributed, then a parametric method (t test) will be used for analysis, otherwise a non-parametric or semi-parametric method will be used (0.5 quantile [median] regression for non-time-to-event data and Cox regression for time-to-event data). Data will be presented as mean, SD (standard deviation) (for normally-distributed outcomes) or median/ IQR (interquartile range) (for non-normally-distributed outcomes). 95% CIs for the differences between groups will be constructed using standard techniques (for normally-distributed outcomes) or using bootstrapping of 10,000 replications (for non-normally-distributed outcomes).

Categorical outcomes will be analyzed using Fisher's exact test, along with the relative risk and its two-sided 95% CI (confidence interval).

Regression adjustment will be performed for any prognostically-important differences between groups in baseline variables.

A P value of < 0.05 will be considered significant

Randomization and Blinding Participants will be randomized to one of two groups by a computer-generated sequence using Lawson Redcap by one of the study members. The investigators, participants, and outcome assessors will be blinded to participant group assignment at the time of randomization as well as throughout treatment and assessment. The drugs will be prepared by one of the study members who will not be involved directly in the patient's care that day.

Data Collection Data will be collected on case record forms. Each form will be signed and dated by the assessor. Paper files will be stored in the locked office of the study PI in the Anesthesia Department at Victoria Hospital, LHSC. Electronic data will be kept in the REDCap database which is housed with the Lawson Research Informatics servers in the hospital's data centre Collection

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective VATS lung resections including wedge resection, segmentectomy, bi-lobectomy, or lobectomy.
* Age > 18 years.
* ASA (American Society of Anesthesiology) Score - 1 to 4.
* Gender - all genders
* Patients able to consent to participate in the study

Exclusion Criteria:

* Patient refusal to participate in the study.
* Emergency surgery.
* Allergies to local anesthetics
* BMI>40
* Presence of local (chest wall) or systemic infection.
* Previous lung resection on the same hemithorax.
* Patient suffering from chronic pain defined by persistent pain more than six month.
* Conversion to thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | Measured on postoperative day 1
  Measured using the Quality of Recovery 40 (Qor-40) Score and asking patients to complete the questions.

SECONDARY OUTCOMES:
Postoperative pain scores | Until patient discharge, on average one week.
  Pain will be assessed on an 11- point numerical scale of '0' to '10'. Zero signifies no pain whereas 10 signifies maximum pain. Measured by asking patient to rate their pain using this scale. This will be measured every 24 hours following surgery until the patient is discharged, on average one week.
Total opioid consumption | Until patient discharge, on average one week.
  Total opioid consumption will be administered in IV morphine equivalents. This will be assessed daily upon admission to post-anesthesia care unit (postoperative care unit) until day of discharge, on average one week. Measured by evaluating patient's medical record for administered morphine equivalents.
Postoperative complications after thoracic surgery | Immediately following surgery until discharge, on average one week.
  Any complication that requires assessment and/or treatment postoperatively. This will be recorded by evaluating the patient's medical chart for any noted complication following surgery.
Hospital readmission | 30 days postoperative
  Instances that the patient may be re-admitted to the hospital following discharge after surgery. To be measured by evaluating the patient's medical record.
Side effects | Until patient discharge, on average one week.
  Side effects will be recorded only if the patient has received an intervention and needed treatment. This will be measured by asking patients each day whether or not they are experiencing any side effects. Patients complaining of mild side effects, like nausea, pruritus or retention of urine, had these effects resolved without administration of any treatment inform of medication or interventions like catheterisation, will be not be counted for this study purpose. Side effects include: nausea and vomiting (needing medication for treatment), pruritus (needing medication for treatment), and retention of urine needing catheterization. This will be measured by recording the type of side effect experienced and the frequency with which the patient mentioned experiencing them.

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Biswas, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontairo, Canada

IPD SHARING:
Plan to Share IPD: No
None. No plan to share IPD (individual participant data).

REFERENCES:
- [Background] Agostini P, Lugg ST, Adams K, Vartsaba N, Kalkat MS, Rajesh PB, Steyn RS, Naidu B, Rushton A, Bishay E. Postoperative pulmonary complications and rehabilitation requirements following lobectomy: a propensity score matched study of patients undergoing video-assisted thoracoscopic surgery versus thoracotomydagger. Interact Cardiovasc Thorac Surg. 2017 Jun 1;24(6):931-937. doi: 10.1093/icvts/ivx002. PMID 28329213
- [Background] Horno Gonzalez R, Gomez-Arnau J, Garcia de Sola R, Arcas M, Avello Garcia F. [Anesthetic management in dorsal rhizotomy by selective cryotherapy and percutaneous thermocoagulation]. Rev Esp Anestesiol Reanim. 1981 Nov;28(6):326-8. No abstract available. Spanish. PMID 7330380
- [Background] Cattaneo SM, Park BJ, Wilton AS, Seshan VE, Bains MS, Downey RJ, Flores RM, Rizk N, Rusch VW. Use of video-assisted thoracic surgery for lobectomy in the elderly results in fewer complications. Ann Thorac Surg. 2008 Jan;85(1):231-5; discussion 235-6. doi: 10.1016/j.athoracsur.2007.07.080. PMID 18154816
- [Background] Marshall K, McLaughlin K. Pain Management in Thoracic Surgery. Thorac Surg Clin. 2020 Aug;30(3):339-346. doi: 10.1016/j.thorsurg.2020.03.001. Epub 2020 Apr 29. PMID 32593366
- [Background] Heinrich S, Janitz K, Merkel S, Klein P, Schmidt J. Short- and long term effects of epidural analgesia on morbidity and mortality of esophageal cancer surgery. Langenbecks Arch Surg. 2015 Jan;400(1):19-26. doi: 10.1007/s00423-014-1248-9. Epub 2014 Sep 21. PMID 25240610
- [Background] Saeki H, Ishimura H, Higashi H, Kitagawa D, Tanaka J, Maruyama R, Katoh H, Shimazoe H, Yamauchi K, Ayabe H, Kakeji Y, Morita M, Maehara Y. Postoperative management using intensive patient-controlled epidural analgesia and early rehabilitation after an esophagectomy. Surg Today. 2009;39(6):476-80. doi: 10.1007/s00595-008-3924-2. Epub 2009 May 27. PMID 19468802
- [Background] LHSC, data support team financial year 2017-2018
- [Background] Bernhard GC. Auranofin treatment for adult rheumatoid arthritis. Comparison of 2 mg and 6 mg daily dose. J Rheumatol Suppl. 1982 Jul-Aug;8:149-53. PMID 6813477
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795
- [Background] Hermanides J, Hollmann MW, Stevens MF, Lirk P. Failed epidural: causes and management. Br J Anaesth. 2012 Aug;109(2):144-54. doi: 10.1093/bja/aes214. Epub 2012 Jun 26. PMID 22735301
- [Background] McLeod G, Davies H, Munnoch N, Bannister J, MacRae W. Postoperative pain relief using thoracic epidural analgesia: outstanding success and disappointing failures. Anaesthesia. 2001 Jan;56(1):75-81. doi: 10.1046/j.1365-2044.2001.01763-7.x. PMID 11167441
- [Background] Naja Z, Lonnqvist PA. Somatic paravertebral nerve blockade. Incidence of failed block and complications. Anaesthesia. 2001 Dec;56(12):1184-8. doi: 10.1046/j.1365-2044.2001.02084-2.x. PMID 11736777
- [Background] Snyder S. Isolated sleep paralysis after rapid time-zone change ('jet-lag') syndrome. Chronobiologia. 1983 Oct-Dec;10(4):377-9. No abstract available. PMID 6661984
- [Background] Viti A, Bertoglio P, Zamperini M, Tubaro A, Menestrina N, Bonadiman S, Avesani R, Guerriero M, Terzi A. Serratus plane block for video-assisted thoracoscopic surgery major lung resection: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2020 Mar 1;30(3):366-372. doi: 10.1093/icvts/ivz289. PMID 31808538
- [Background] Kim DH, Oh YJ, Lee JG, Ha D, Chang YJ, Kwak HJ. Efficacy of Ultrasound-Guided Serratus Plane Block on Postoperative Quality of Recovery and Analgesia After Video-Assisted Thoracic Surgery: A Randomized, Triple-Blind, Placebo-Controlled Study. Anesth Analg. 2018 Apr;126(4):1353-1361. doi: 10.1213/ANE.0000000000002779. PMID 29324496
- [Background] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Background] Kain ZN, Vakharia S, Garson L, Engwall S, Schwarzkopf R, Gupta R, Cannesson M. The perioperative surgical home as a future perioperative practice model. Anesth Analg. 2014 May;118(5):1126-30. doi: 10.1213/ANE.0000000000000190. No abstract available. PMID 24781578
- [Background] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540